CLINICAL TRIAL: NCT04337788
Title: Gerontological Telemonitoring of Older Adults Living in Nursing Homes With Symptoms of Confirmed or Probable COVID-19 Disease
Brief Title: Gerontological Telemonitoring of Older Adults Living in Nursing Homes With COVID-19 Disease
Acronym: COVIDeHPAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 87RI20_0013
Record Dates: First submitted 2020-04-03; First posted 2020-04-08 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-04

CONDITIONS: Coronavirus Infection
Keywords: Covid-19, early gerontologic healthcare
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Intervention Model Description: Prospective cohort study (here and elsewhere)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- gerontological telemonitoring action (Experimental): Nurses answer a daily resident-reported questionnaire (e.g. temperature, dyspnea, pain), edited by French health authorities. From D0 to D20, data are transmitted to the NHSP. Warning algorithms specially developed for older persons identify signs that are monitored by the NHSP geriatrician coordinator. A feedback is provided to the general physician for specific actions required and appropriate support.
  A last questionnaire is completed at D30 by the nurse in order to stop monitoring and know event occurred between D20 to D30.
  Interventions: Other: telehealth applications
- routine care without gerontological telemonitoring (No Intervention): routine care

INTERVENTIONS:
Other: telehealth applications — telehealth applications during 30 days/patient
  Arms: gerontological telemonitoring action

SUMMARY:
Since the last 3 months the world copes with the novel coronavirus disease : Covid-19 emerged in China in the end of 2019. WHO declared the pandemic situation as a Public Health Emergency around the world on January 2020.

Firsts studies emphasized on higher risk to older adults to experience serious health consequences : hospitalizations and mortality, due to multimorbidity and multimedication. Nursing home resident are particulary frailer and vulnerable.

ELIGIBILITY:
Inclusion Criteria:

* Nursing home resident with Covid disease RT-PCR or Chest CT or rapid test
* Nursing home resident with Covid-19 disease symptoms :
* fever
* cough
* dyspnea
* SPO2<95% in ambient air (or <91% in COPD patient)
* Diarrhea
* Fall or balance disorder
* Confusion

Exclusion Criteria:

* Age < 75 years
* Patient in respiratory distress
* No consent

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-05 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Impact of Gerontological telemonitoring on healthcare management for older adults living in Nursing Homes with symptoms of confirmed or probable COVID-19 disease (Death within 30 days). | day 30

IPD SHARING:
Plan to Share IPD: No